CLINICAL TRIAL: NCT01503970
Title: Autologous Chondrocyte Transplantation For Articular Cartilage Regeneration. Pilot Study
Brief Title: Autologous Chondrocyte Transplantation For Articular Cartilage Regeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Aldo Izaguirre, Study Director, Instituto Nacional de Rehabilitacion
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 017-04-INR
Record Dates: First submitted 2011-12-01; First posted 2012-01-04 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Tear; Knee, Cartilage, Articular
Keywords: chondral lesions; knee
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chondrocyte implantation (Experimental)
  Interventions: Device: Arthroscopic matrix encapsulated chondrocyte implantation

INTERVENTIONS:
Device: Arthroscopic matrix encapsulated chondrocyte implantation — Each implant of collagen scaffold contains approximately 6,000,000 autologous chondrocytes. This constructs of 10 mm diameter are implanted arthroscopically at the defect.

SUMMARY:
The purpose of this study is to assess safety and efficacy of autologous chondrocyte implantation delivered arthroscopically into chondral lesions of the knee using clinical, biochemical, and MRI outcomes.

DETAILED DESCRIPTION:
Injuries to the articular cartilage of the knee are common. They produce pain and deteriotation of patients' quality of life. The management of focal chondral lesions continues to be problematic for the treating orthopaedic surgeon. Although many treatment options are currently available, none fulfill the criteria for an ideal repair solution: a hyaline repair tissue that completely fills the defect and integrates well with the surrounding normal cartilage. Autologous chondrocyte implantation is a relatively new cell-based treatment method for full-thickness cartilage injuries that in recent years has increased in popularity, with different studies showing promising results. Typically, this implantation is performed in an open-surgery fashion. In our study the implantation of in-house autologous chondrocyte culture is done arthroscopically, situation that may offer advantages in surgery associated morbidity and patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic chondral lesions of the knee

Exclusion Criteria:

* Inflammatory arthritis
* Septic arthritis
* Total meniscectomy
* Previous microfracture at chondral lesions
* Paget
* Ochronosis
* Acromegalia

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to different periods in T2 Mapping for cartilage lesions after treatment. | 3, 6, 9, 12, 18, 24 36 months
  Special magnetic resonance imaging technique for measurement of collagen and water content, it is expressed in milliseconds.

SECONDARY OUTCOMES:
Change of baseline to different periods in Clinical evaluation | 0, 10, 30 days, 3, 6, 9, 12, 24, 36 months
  Clinical assessment with validated knee scores, and adverse effects register are taken.

CONTACTS AND LOCATIONS:
Overall Officials: Clemente Ibarra, M.D., Principal Investigator — INR; Luis Guillermo Ibarra, M.D., Study Chair — INR; Aldo F Izaguirre, M.D., Study Director — INR; Enrique Villalobos, M.D., Study Director — INR
Locations (1):
- National Rehabilitation Institute, Mexico City, Mexico

REFERENCES:
- [Background] Masri M, Lombardero G, Velasquillo C, Martinez V, Neri R, Villegas H, Ibarra C. Matrix-encapsulation cell-seeding technique to prevent cell detachment during arthroscopic implantation of matrix-induced autologous chondrocytes. Arthroscopy. 2007 Aug;23(8):877-83. doi: 10.1016/j.arthro.2007.05.010. PMID 17681210
- [Background] Ibarra-Ponce de Leon JC, Velasquillo-Martinez MC, Izaguirre A, Villalobos-Cordova E, Masri M, Ibarra-Ibarra LG. [Cartilage repair: cell-based techniques]. Acta Ortop Mex. 2009 Jan-Feb;23(1):38-44. Spanish. PMID 19462773
- [Background] Ibarra C, Izaguirre A, Villalobos E, Masri M, Lombardero G, Martinez V, Velasquillo C, Meza AO, Guevara V, Ibarra LG. Follow-up of a new arthroscopic technique for implantation of matrix-encapsulated autologous chondrocytes in the knee. Arthroscopy. 2014 Jun;30(6):715-23. doi: 10.1016/j.arthro.2014.02.032. Epub 2014 Apr 18. PMID 24746406